CLINICAL TRIAL: NCT07008144
Title: Introducing Electronic Alerts to Reduce Inappropriate Digoxin Prescribing in Older Adults
Acronym: Aldigo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CSAPG-73
Record Dates: First submitted 2025-05-26; First posted 2025-06-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Drug-Related Side Effects and Adverse Reaction; Digoxin Overdose
Keywords: digoxin; deprescription; Beers; computerized alerts; geriatrics; Elderly Hospitalized Patients
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Before intervention (No Intervention): In this group, the outcome will be measured before the intervention is implemented at the center
- Post intervention (Experimental): In this group, the outcome will be measured after the intervention is implemented at the center
  Interventions: Other: Digoxin alarm

INTERVENTIONS:
Other: Digoxin alarm — A computerized alert will be integrated into the CSAPG electronic health record system (MIRA software). These alerts will be triggered when a physician prescribes digoxin at a dose higher than the recommended 0.125 mg/day for elderly patients.
  Arms: Post intervention

SUMMARY:
The intervention consists of introducing computerized alerts into the electronic medical record of the CSAPG (MIRA software), which are triggered when a physician prescribes digoxin at a dose higher than the recommended amount (more than 0.125 mg/day).

The main objective of this study is to evaluate the effectiveness of a visible computerized alert aimed at physicians responsible for hospitalized elderly patients who have been prescribed digoxin at a dose higher than 0.125 mg/day (the recommended dose), in reducing the number of patients receiving inappropriate digoxin doses.

DETAILED DESCRIPTION:
Intervention This quasi-experimental pre-post intervention study evaluates the effectiveness of computerized alerts integrated into the CSAPG electronic health record system (MIRA software). These alerts are triggered when a physician prescribes digoxin at a dose higher than the recommended 0.125 mg/day for elderly patients.

Study Objective The main goal is to assess whether these alerts reduce the number of elderly hospitalized patients receiving inappropriate digoxin dosages.

Study Design and Duration The study will last 18 months in total, with a 12-month data collection period at each site (6 months before and 6 months after the intervention).

Sample Size and Population To detect a 25% reduction in inappropriate digoxin prescriptions with 80% power and a 0.05 alpha risk, the study requires 2,977 patients in both the pre- and post-intervention groups. Inclusion criteria include hospitalized men and women aged 65 and older. No patient exclusions are anticipated.

Statistical Analysis The primary analysis will compare the proportion of patients receiving digoxin doses above the recommended level before and after the intervention using the Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 64 years of age.
* Hospitalized in inpatient wards of the study centers during the study period.

Exclusion Criteria:

* Pacients under 64 years old
* Patients without complete data available

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5954 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of elderly inpatients receiving inappropriate digoxin doses | From baseline to hospital discharge, as much 3 months
  Proportion of patients aged 65 and older who are prescribed digoxin at a dose higher than 0.125 mg/day during hospitalization. The outcome compares this proportion between the pre-intervention and post-intervention periods to evaluate the effectiveness of a computerized alert integrated into the electronic medical record system (MIRA).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Rodríguez Molinero, Study Director — Consorci Sanitari de l'Alt Penedès i Garraf
Locations (2):
- Spain (2):
  - Consorci Sanitari Alt Penedès-Garraf-Hospital de Vilafranca, Vilafranca del Penedès, Barcelona
  - Consorci Sanitari Alt Penedès-Garraf Hospital Sant Camil, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.